CLINICAL TRIAL: NCT00264563
Title: "Iatrogenesis Imperfecta"- Extent and Characteristic in NICU in Israel.
Status: Completed | Type: Observational
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Amir Kugelman, Bnai Zion Medical Center
Other Study IDs: 80/05
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2005-08

CONDITIONS: Iatrogenesis in NICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Behavioral: The intervention is basically by letting the care givers to be aware that there is active recording of iatrogenesis
  Interventions: Behavioral: Increasing the level of awareness to Iatrogenesis; Behavioral: Increasing awareness .

INTERVENTIONS:
Behavioral: Increasing the level of awareness to Iatrogenesis — Increasing the level of awareness to Iatrogenesis
Behavioral: Increasing awareness . — Increasing awareness to Iatrogenesis and active daily recordings
  Other Names: In the first 3 months the medical teams were unaware of recordings while in next 3 months they became aware to recordings

SUMMARY:
Iatrogenesis is inevitable in the NICUs.

DETAILED DESCRIPTION:
In the first 3 months of the study we will document Iatrogenic events in 3 NICUs in Israel without informing the medical and nursing staff. In the second 3 months of the study we will try to draw the attention of the medical and nursing staff that we are documenting iatogenesis, and we will assess wether this intervention will decrease the events of Iatrogenesis.

ELIGIBILITY:
Inclusion Criteria:All infants in NICU -

Exclusion Criteria:None

-

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Ifants admitted to NICU during the study period
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2005-11; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Overall Officials: Amir Kugelman, Principal Investigator — Senior Neonatologist
Locations (2):
- Israel (2):
  - Bnai Zion Medical Center, Haifa
  - Bnai Zion Medical Center, Rambam Medical Center, Barzilay Medical Center, Haifa Ans Ashkelon